CLINICAL TRIAL: NCT05263609
Title: Optimizing Pembrolizumab Therapy With Timing and Intensification With Axitinib in Metastatic Renal Cell Cancer: A Response Adapted Study (OPTIMAX)
Brief Title: Optimizing Pembrolizumab Therapy With Timing and Intensification With Axitinib
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI left University
Sponsor: University of Oklahoma (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OU-SCC-OPTIMAX
Record Dates: First submitted 2022-01-24; First posted 2022-03-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Renal Cell Cancer
Keywords: axitinib; pembrolizumab; metastatic renal cell cancer; renal cell cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Arm A (CR/oPR on pembrolizumab monotherapy):
  Patients will continue pembrolizumab monotherapy if CR/oPR on initial treatment with pembrolizumab monotherapy. If CR/oPR persists at 8 cycles (24 weeks) after assignment on arm A, pembrolizumab break will commence. Patients will be monitored for disease progression with imaging every 9 weeks (+/- 1 week). If patients develop progression, pembrolizumab will be resumed and continued until subsequent PD. At that point, axitinib may be added to pembrolizumab as part of the study or patients may discontinue study treatment per the treating investigator's discretion.
  Interventions: Drug: Pembrolizumab
- Arm B (Experimental): Arm B (sPR/SD/PD):
  Patients with sPR, SD or PD after 6 cycles of pembrolizumab monotherapy will be started on axitinib in addition to continuing pembrolizumab. If patients develop subsequent PD, treatment will be discontinued. If the subsequent scans show SD/PR/CR, the combination treatment will be continued until PD or unacceptable toxicity.
  Interventions: Drug: Axitinib

INTERVENTIONS:
Drug: Axitinib — If pembrolizumab infusions alone do not reduce the patient's tumor size by at least 60%,the patient will be placed in Arm B and start axitinib in addition to continuing pembrolizumab therapy (see Arm B).
  Arms: Arm B
Drug: Pembrolizumab — If pembrolizumab results in a reduction in tumor size that is greater than 60%, the patient will be placed in Arm A and continue pembrolizumab infusions (see Arm A).
  Arms: Arm A

SUMMARY:
The purpose of this research is to test the response of study participants' tumor to pembrolizumab alone, and in combination with axitinib, and to see what effects (good and bad) these drugs have on patients with advanced kidney cancer.

DETAILED DESCRIPTION:
Patients will receive infusions of pembrolizumab. After an MRI or CT scan to determine how the tumor is responding to the drug, the patient will either continue receiving infusions of pembrolizumab alone, or receive axitinib in addition to pembrolizumab. The patient will also need to provide a biopsy of your tumor around the time the imaging scan is taken and need to come to the clinic around every three weeks during treatment. At the clinic visits, we will also do lab tests and imaging.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of consent.
* ECOG performance status ≤1 (Appendix A) within 28 days prior to registration.
* Participants must have histologically or cytologically confirmed clear-cell or non-clear cell renal cell carcinoma.
* Presence of measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.137.
* Both previously untreated and treated patients will be eligible for participation with no limit on number of prior lines of therapy. Prior therapy with checkpoint inhibitors and/or axitinib for advanced disease is not allowed. Patients who have received treatment with prior checkpoint inhibitors (anti-PD-1/L1 or anti- CTLA-4) or VEGF receptor tyrosine kinase inhibitors in neoadjuvant/adjuvant setting are eligible for inclusion if time from treatment discontinuation to disease recurrence is more than 1 year.
* Adequately controlled blood pressure (BP), with or without antihypertensive medications, defined as BP ≤150/90 mmHg at screening and no change in antihypertensive medications within 1 week before the Cycle 1/Day 1.
* Willingness of the patient to undergo mandatory fresh tumor biopsy on study unless determined medically unsafe or not feasible by the treating investigator. If a target lesion is biopsied at screening, this lesion must be followed as non-target lesion after the biopsy unless it is the patient's only target lesion.
* Participants must have normal organ and marrow function as defined below within 42 days prior to first study treatment
* A female participant is eligible to participate if they are not pregnant (negative urine or serum pregnancy test within 42 days prior to registration), not breastfeeding, and at least one of the following conditions applies: a.) Not a woman of childbearing potential (WOCBP) OR b.) A WOCBP who agrees to follow tcontraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.
* A male participant must agree to use contraception as of this protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.

Exclusion Criteria:

* Participants who have had prior systemic checkpoint inhibitors (anti-PD-1/L1 or anti-CTLA-4) and/or axitinib for the management of metastatic RCC.
* Participants who have had any type of anti-cancer therapy (including investigational therapy, monoclonal antibodies, cytokine therapy, small molecule kinase inhibitor or chemotherapy) within 2 weeks prior to enrollment on the study.
* Radiotherapy for RCC within 14 days of first study treatment with the exception of a single fraction of radiation administered for palliation of symptoms.
* Presence of any toxicities attributed to prior anti-cancer therapy that are not resolved to ≤ grade 1 (National Cancer Institute Common Terminology Criteria for Adverse Events CTCAE version v5.0) or baseline before administration of study drug38 with the exception of alopecia or grade 2 fatigue.
* Participants who are receiving systemic immunosuppressive medications within 2 weeks of first study dose, including but not limited to: prednisone, dexamethasone, cyclosporin, azathioprine, methotrexate, thalidomide, anti-tumor necrosis factor (TNF) agents
* Treatment with short term (<7 days), or low-dose systemic immunosuppressant medications (≤ 10 mg prednisone/day equivalent) within 2 weeks of first study dose is permitted.
* Patients with adrenal insufficiency on physiologic replacement doses of steroids (≤ 10 mg prednisone equivalent) may be enrolled.
* The use of inhaled, topical, ocular or intra-articular corticosteroids and mineralocorticoids are allowed for other non-RCC co-morbidities.
* Any active or recent history (within 6 months of first study dose) of autoimmune disease or syndrome that requires systemic corticosteroids (>10 mg daily prednisone equivalent) or immunosuppressive medications.
* Patients with low risk disorders, such as vitiligo, controlled type I diabetes mellitus, hypo- or hyperthyroid disease, or surgical adrenal insufficiency requiring hormone replacement therapy, are permitted to enroll. Discuss with PI any additional disorders not on this list that may qualify.
* Participants with known untreated or symptomatic metastases to the brain, spinal cord or leptomeninges. Patients may be eligible if stable intracranial disease for at least 4 weeks before first study treatment as documented by magnetic resonance imaging (MRI) or computerized tomography (CT) imaging and if no ongoing requirement for steroids.
* Prolonged corrected QT interval by the Fridericia correction formula (QTcF) on screening ECG > 480 msec.
* Bleeding or thrombotic disorders or patients at risk for severe hemorrhage. Gastrointestinal malabsorption, gastrointestinal anastomosis, fistula, or any other condition that might affect the absorption of axitinib.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab or axitinib.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Known active or chronic hepatitis B infection (defined as having a positive hepatitis B surface antigen (HBsAg) test at screening).
* Patient with past or resolved hepatitis B infection (defined as having a negative HBsAg test and positive antibody to hepatitis B core antigen test) are eligible. Hepatitis B viral DNA must be obtained in patients with positive hepatitis B core antibody prior to first treatment start.
* Patients with active/chronic viral hepatitis C are ineligible because of the potential for pharmacokinetic interactions.
* Patients with positive hepatitis C antibody test are eligible if PCR is negative for hepatitis C viral DNA.
* Known HIV-positive participants are ineligible because of the potential for pharmacokinetic interactions and an increased risk of lethal infections when treated with immunosuppressive therapy for immune related adverse events.
* Administration of a live vaccine or live-attenuated vaccine within 30 days of first dose of study treatment. Administration of killed vaccine is allowed.
* Receipt of therapeutic oral or IV antibiotics within 2 weeks of first study treatment. Patients receiving routine antibiotic prophylaxis (for dental extractions/procedures) are eligible. Empiric antibiotics given without subsequent proof of infection will not be counted as ineligible.
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Prior allogenic stem cell or solid organ transplant.
* Other malignancies with the exception of those with negligible risk of metastases or death in view of the treating investigator and/or treated with expected curative outcome. Examples of (but not limited to) permitted treated cancers: carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, ductal carcinoma in situ of the breast, non-muscle invasive urothelial carcinoma not requiring current therapy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patient Response | 2 year
  To catalogue the number and proportion of patients with persistence of complete response or optimal partial response at 1 year after the discontinuation of pembrolizumab
Objective Response Rate After Axitinib | 2 year
  To assess the objective response rate after addition of axitinib in patients with a suboptimal partial response, stable disease or progressive disease on pembrolizumab monotherapy alone.

SECONDARY OUTCOMES:
Objective Response Rate after Pembrolizumab | 2 year
  To determine the objective response rate (ORR: CR +oPR + sPR) after 6 cycles of primary treatment with pembrolizumab
Duration of Response | 2 year
  To determine duration of CR or oPR
  To determine progression-free survival (PFS) from pembrolizumab initiation
  To determine treatment-free survival (TFS) from pembrolizumab discontinuation
  To assess safety and toxicity according to NCI CTCAE v5
Overall Survival | 2 year
  To determine overall survival (OS) from pembrolizumab initiation
Proportion of patients that experience toxicity | 2 year
  To assess safety and toxicity according to NCI CTCAE v5 on pembrolizumab monotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Tripathi, MD, Principal Investigator — Stephenson Cancer Center

IPD SHARING:
Plan to Share IPD: No